CLINICAL TRIAL: NCT02056977
Title: Comparison Between PEEP Levels Selected by Individualized PEEP Titration - Rapid Titration by EIT - and PEEP Levels Routinely Used in Post-operative Cardiac Patients With Hypoxemic Respiratory Failure
Brief Title: PEEP Levels Selected by PEEP Titration and PEEP Levels Routinely Used in Post-operative Cardiac Patients With Hypoxemic Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 513.205
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Post Operative Cardiac Surgery; ARDS; Hypoxemic Respiratory Failure
Keywords: Acute Respiratory Distress Syndrome; Cardiac Surgical Procedure; Mechanical Ventilation; Postoperative Complications; Positive End-Expiratory Pressure; Lung Collapse; Respiratory Failure; Electrical Impedance Tomography
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Postoperative Complications; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Titration (Experimental): Individualized PEEP titration by EIT
  Interventions: Other: Titration
- Control (Active Comparator): PEEP stablished according to the routines at the institution (PEEP table according to the P/F ratio)
  Interventions: Other: control

INTERVENTIONS:
Other: Titration — Individualized PEEP according to PEEP titration monitored by EIT
  Other Names: Individualized PEEP
  Arms: Titration
Other: control — PEEP selected according to a PaO2/FIO2 table as in the routines of the institution
  Other Names: Control PEEP
  Arms: Control

SUMMARY:
The purpose of this study is to:

* Compare PEEP level selected by individualized PEEP titration by electrical impedance tomography and PEEP level routinely used in post-operative cardiac patients with Hypoxemic Respiratory Failure;
* Evaluate the agreement between the results of a rapid titration (total procedure duration = 5 min) versus an already validated slow titration (total procedure duration = 40 min) of the same patient, sequentially. Specifically, degree of collapse and degree of distention in each PEEP level, estimated by EIT;
* Compare hemodynamics during the two maneuvers of PEEP titration;
* Evaluate the efficacy of the selected PEEP (minimum PEEP preventing lung collapse less than 5%) to maintain stable levels of the following variables: arterial oxygenation, respiratory system compliance, and degree of collapse by EIT;
* Compare these results (evolution of the three variables, along 4 hours) with the control strategy (default strategy currently used in the institution) group.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) increases the morbidity and mortality of patients admitted to the intensive care unit (ICU). In the postoperative period of cardiac surgery, the use of intraoperative extracorporeal circulation is one of the factors triggering the syndrome, its incidence increasing.

Potentially, a protective ventilatory strategy with optimal positive end expiratory pressure (PEEP) could improve the prognosis of those patients with ARDS.

An already validated maneuver to titrate the ideal PEEP to these patients has a longer duration, about 40 minutes. The lung Electrical impedance tomography (EIT) monitors respiratory system mechanics and intrathoracic lung volume changes and provides information about regional behavior and recruitability of lung tissue and thereby allows shortening titration maneuver, reducing its hemodynamic effects.

Patients in the postoperative period of cardiac surgery with a diagnosis of Hypoxemic Respiratory Failure (PaO2/FiO2 < 250 mmHg, calculated at FiO2 60%, and the presence of bilateral infiltrates on chest radiography), admitted to the surgical ICU from Heart Institute, University of São Paulo.

Recruitment maneuver and PEEP titration maneuver will be monitored by EIT.

All patients will be followed and monitored for 4 hours, with measures of the evolution of alveolar collapse . Hemodynamic and oxygenation data will also be recorded .

ELIGIBILITY:
Inclusion Criteria:

* Immediate postoperative period of myocardial revascularization and/or heart valve surgery (aortic and/or mitral)
* Acute respiratory distress syndrome with ratio of partial pressure of arterial oxygen over fraction of inspired oxygen (PaO2:FiO2) no >200 mmHg and bilateral pulmonary infiltrates on XRay consistent with edema, and no clinical evidence of left atrial hypertension (pulmonary capillary wedge pressure <18 mmHg, when available).
* Age > 18 and < 70 years old
* Absence previous pulmonary disease
* Left ventricular ejection fraction > 35%
* Absence of previous cardiac surgery and / or lung disease;
* Not requiring adjusted volume expansion (pulse pressure delta <13% or legs raising test without hemodynamic changes in cardiac index or mean arterial pressure).
* Body mass index < 40 kg/m2
* Written inform consent

Exclusion Criteria:

* MAP < 70 mmHg
* Noradrenaline > 1 micrograms/Kg/min
* Acute arrhythmias
* Blooding associated to hemodynamic instability
* Need of re-surgery and/or mechanical circulatory assistance
* Suspicion of neurological alteration
* Chest tube with persistent air leak

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
To test the agreement between the ideal PEEP determined by rapid titration versus and the ideal PEEP determined by the slow PEEP titration maneuver. | 2 hours
  Evaluate the agreement between the ideal PEEP determined by the rapid PEEP titration maneuver versus the ideal PEEP determined by the slow PEEP titration maneuver. The degree of collapse and overdistention at each PEEP level, as estimated by EIT, will be also compared during both procedures. Ideal PEEP is the minimum PEEP capable of keeping collapse at < 5%.

SECONDARY OUTCOMES:
Stability of the selected PEEP according to the rapid titration in arterial oxygenation (SpO2, in %), respiratory system compliance (in cmH2O), and degree of collapse by EIT (in %) | 4 hours
  Evaluate the stability of the selected PEEP (according to the rapid titration), by analyzing the maintenance of three variables over a four hour period: arterial oxygenation, respiratory system compliance, and degree of collapse by EIT

OTHER OUTCOMES:
Comparison of the PEEP levels selected by the proposed strategy (rapid titration maneuver) and the PEEP levels used in the control group. | 4 hours
  To compare the values of PEEP selected by both strategies, and to compare the evolution of the three variables (arterial oxygenation, respiratory system compliance, and degree of collapse by EIT) between propose strategy to control (default strategy currently used in the institution)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo BP Amato, Principal Investigator — Department of Cardio-Pulmonar, Pulmonary Division, Hospital das Clínicas, University of São Paulo
Locations (1):
- USP Instituto do Coração, São Paulo, Brazil

REFERENCES:
- [Background] Costa EL, Amato M. Hemodynamic and respiratory changes during lung recruitment and descending optimal positive end-expiratory pressure titration with acute respiratory distress syndrome. Crit Care Med. 2007 Aug;35(8):1998-9; author reply 1999. doi: 10.1097/01.ccm.0000277060.87425.6b. No abstract available. PMID 17667256